CLINICAL TRIAL: NCT06908811
Title: Effect of a Novel Blend of Plant Protein and Additional Ingredients on Resistance Training Adaptations
Acronym: IOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB-22-67
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Resistance Exercise
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Parallel Design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Supplements were blinded, in labeled containers. Each supplement will be of a similar volume, texture, and flavor, and labeled in indistinguishable packaging to ensure blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Novel Plant Protein (Experimental): Novel plant protein blend containing 30 grams of protein taken twice per day for 8 weeks
  Interventions: Dietary Supplement: Novel Plant Protein Blend
- Pea/Rice Protein (Active Comparator): Pea/Rice protein blend containing 30 grams of protein taken twice per day for 8 weeks
  Interventions: Dietary Supplement: Pea/Rice Protein Blend
- Whey Protein (Active Comparator): Whey protein blend containing 30 grams of protein taken twice per day for 8 weeks
  Interventions: Dietary Supplement: Whey Protein
- Carbohydrate Placebo (Placebo Comparator): Carbohydrate placebo (maltodextrin) taken twice per day for 8 weeks
  Interventions: Dietary Supplement: Carbohydrate Placebo

INTERVENTIONS:
Dietary Supplement: Novel Plant Protein Blend — Novel plant protein blend containing 30 grams of protein.
  Arms: Novel Plant Protein
Dietary Supplement: Pea/Rice Protein Blend — Pea/Rice protein blend containing 30 grams of protein
  Arms: Pea/Rice Protein
Dietary Supplement: Whey Protein — Whey concentrate protein blend containing 30 grams of protein
  Arms: Whey Protein
Dietary Supplement: Carbohydrate Placebo — Maltodextrin placebo
  Arms: Carbohydrate Placebo

SUMMARY:
This study seeks to compare the observed changes in resistance training adaptations (strength, performance, body composition, recovery, and lactate responses) after supplementation of isocaloric and isonitrogenous amounts of a novel plant protein formulation against changes observed in a pea/rice plant protein blend, whey protein, and a carbohydrate placebo in healthy resistance-trained men and women between the ages of 18-39.

DETAILED DESCRIPTION:
This study seeks to compare the observed changes in resistance training adaptations (strength, performance, body composition, recovery, and lactate responses) after supplementation of isocaloric and isonitrogenous amounts of a novel plant protein formulation against changes observed in a pea/rice plant protein blend, whey protein, and a carbohydrate placebo in healthy resistance-trained men and women between the ages of 18-39.

ELIGIBILITY:
Inclusion Criteria

* Between the ages of 18-39 years
* Participants will be healthy and free of disease as determined by evaluation of a medical history
* All participants will be required to abstain from taking any additional forms of nutritional supplementation deemed to be ergogenic or that will impact resistance training adaptations (pre-workouts, creatine, beta-alanine, etc.) for four weeks prior to beginning this study and for the entire duration of the study.

Exclusion Criteria

* Those individuals less than 18 and greater than 39 years of age will be excluded.
* Participants who are determined to not be weight stable defined as pre-study and visit 1 body mass levels deviating by 3% or more.
* Any individual who is currently being treated for or diagnosed with a cardiac, respiratory, circulatory, musculoskeletal, metabolic, immune, autoimmune, psychiatric, hematological, neurological or endocrinological disorder or disease.
* Body mass index >29.9 kg/m2. Males with a body mass index greater than 29.9 kg/m2, but a body fat percentage less than 27.5% fat will be accepted into the study. Females with a body mass index greater than 29.9 kg/m2, but a body fat percentage less than 32.5% fat will be accepted into the study. The average body mass index for the entire study cohort will be less than 27.5 kg/m2. As such, an ongoing calculation of the recruited cohort's mean body mass index will be maintained and people will only be randomized into the study if the average cohort body mass index value does not exceed 27.5 kg/m2
* Individuals who present with any previous injury or illness that would prevent them from appropriately completing all exercise lifts.
* Participants who are not able to fit onto the DEXA table will not be able to participate in the research due to size restrictions of the equipment. This typically includes individuals exceeding 400 pounds or those greater than 6'4".
* Those individuals with less than 3 months of structured resistance training, aerobic training, or team sport participation experience will be excluded from the study.
* Pregnant women, women trying to become pregnant, or nursing women. Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Change in 4-Compartment Lean Mass | Week 0, Week 4, and Week 8
  Lean mass will be assessed using a 4-compartment model, which includes measurements of body density, total body water, and bone mineral content.
Change in Perceptual Indicators of Training State | Week 0, Week 4, and Week 8
  Participants will rate their readiness to train, soreness, recovery, energy, and sleep quality using 100-mm visual analog scales. Each scale is anchored with contextually appropriate statements such as "Lowest Possible" and "Highest Possible."
Change in Profile of Mood States (POMS) Score | Week 0, Week 4, and Week 8
  Mood state will be assessed using the Profile of Mood States (POMS) questionnaire, a validated tool for measuring transient affective states. The POMS consists of six subscales (Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment), with a Total Mood Disturbance (TMD) score calculated by summing negative subscale scores and subtracting the Vigor score. Higher TMD scores indicate greater mood disturbance, while lower scores indicate improved mood state.
Change in Pressure to Pain Threshold | Week 0, Week 4, and Week 8
  Pressure pain threshold will be assessed using a digital algometer to determine the minimum pressure required to elicit pain. Higher scores indicate higher tolerance to pain.
Change in Handgrip Strength | Week 0, Week 4, and Week 8
  Maximal handgrip strength will be assessed using a calibrated hand dynamometer. Higher values indicate greater strength.
Change in Isometric Mid-Thigh Pull Force | Week 0, Week 4, and Week 8
  Maximal force output will be assessed using an isometric mid-thigh pull on a force plate, measured in Newtons. Higher scores equal greater force production
Change in Hex Bar Deadlift One-Repetition Maximum (1RM) | Week 0, Week 4, and Week 8
  Maximal hex bar deadlift strength will be assessed using a standardized one-repetition maximum (1RM) test.
Change in Bench Press One-Repetition Maximum (1RM | Week 0, Week 4, and Week 8
  Maximal upper-body strength will be assessed using a standardized one-repetition maximum (1RM) bench press test.
Change in Isokinetic Peak Knee Extension Torque | Week 0, Week 4, and Week 8
  Peak torque of the quadriceps will be assessed using an isokinetic dynamometer. Higher values indicate greater knee extensor strength.
Performance in 5 Sets of Hex Bar Deadlift Protocol | Week 0, Week 4, and Week 8
  Strength endurance will be assessed using a hex bar deadlift protocol consisting of 3 sets of 10 repetitions at 70% 1RM and 2 sets to failure at 80% 1RM. Repetition count and total volume lifted will be recorded.

SECONDARY OUTCOMES:
Change in 4-Compartment Fat Mass | Week 0, Week 4, and Week 8
  Fat mass will be measured using a 4-compartment model, which integrates body density, total body water, and bone mineral content.
Change in 4-Compartment Fat-Free Mass | Week 0, Week 4, and Week 8
  Fat-free mass will be assessed using a 4-compartment model, providing a more precise measurement of body composition changes.
Change in 4-Compartment Percent Body Fat | Week 0, Week 4, and Week 8
  Body fat percentage will be assessed using a 4-compartment model.
Change in Total, Extracellular, and Intracellular Body Water | Week 0, Week 4, and Week 8
  Hydration status will be measured using bioelectrical impedance analysis (BIA) to assess total, extracellular, and intracellular body water content.
Change in Dry Fat-Free Mass | Week 0, Week 4, and Week 8
  Dry fat-free mass will be assessed using a combination of dual-energy X-ray absorptiometry (DEXA) and bioelectrical impedance analysis (BIA) for a comprehensive measure of lean tissue mass.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared